CLINICAL TRIAL: NCT02208661
Title: Psychological Concomitants of Morquio A Syndrome - Longitudinal Effects of Enzyme Replacement Therapy
Brief Title: Psychological Concomitants of Morquio A Syndrome - Longitudinal Effects of Enzyme Replacement Therapy (The MAPLE Study)
Acronym: MAPLE
Status: Completed | Type: Observational
Sponsor: Nadia Ali, PhD (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor-Investigator, Nadia Ali, PhD, Health Psychologist, Emory University
Organization: Emory University (Other)
Other Study IDs: IRB00072780
Record Dates: First submitted 2014-08-01; First posted 2014-08-05 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Morquio A Syndrome; Mucopolysaccharidosis IV A
Keywords: Morquio A syndrome; Mucopolysaccharidosis IV A; Psychological health
MeSH Terms: conditions — Mucopolysaccharidosis IV; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Mucopolysaccharidosis IV, also known as MPS IV or Morquio disease, is a rare autosomal recessive genetic lysosomal storage disorder. Research thus far regarding Morquio, has primarily focused on the physical aspects of the various diseases. Less attention has been paid to the psychological toll of these diseases, whether they are direct symptoms or reactions to living with a chronic progressive disease.

Prior to 2013, there was neither a cure nor treatment (other than palliative) for Morquio disease. In the latter half of 2013, ERT became available to the broader population of patients with Morquio A disease through BioMarin's Expanded Access Program.

In a previous study, entitled "Psychological Concomitants of Morquio syndrome" the present investigator enrolled 20 adult subjects with Morquio into a pilot study to estimate a baseline incidence of psychological symptoms and overall quality of life. Subjects were all over the age of 18. Data from this study were published in 2015.

The present study extends this research into psychological health with Morquio via a comparison of psychological issues and quality of life before and after treatment (i.e. ERT). As ERT does not cross the blood-brain barrier, it would be unlikely to improve organic psychological symptoms, but may improve any reactive psychological symptoms caused by living over time with this chronic progressive genetic disease.

The present study thus seeks to follow adult patients with Morquio A disease as they begin ERT and track their psychological health every 6 months for a duration of 2 years. Adult patients with Morquio disease are invited to participate. Subjects will complete three different self-report questionnaires, the Achenbach System of Empirically Based Assessment (ASEBA) Adult Self-Report (ASR), the Short Form 36-item Health Questionnaire (SF-36), and the Brief Pain Inventory (BPI). Group aggregate data will be reported; individual questionnaire content and results will be held confidential, except as in accordance with Georgia law relating to reporting of child or elder abuse, suicidal and/or homicidal intent.

DETAILED DESCRIPTION:
Mucopolysaccharidosis IV, also known as MPS IV or Morquio disease, is a rare autosomal recessive genetic lysosomal storage disorder. Research thus far regarding lysosomal storage diseases (LSDs) in general, including Morquio, has primarily focused on exploring the causes of and finding a treatment for the physical aspects of the various diseases. Less attention has been paid to the psychological or emotional toll of these diseases, whether they are direct symptoms of the diseases themselves or reactions to living with a chronic progressive disease.

It is well established in the health psychology literature, however, that the interaction between our physical health and our psychological health is bidirectional; that is, just as our physical health affects us emotionally (e.g. chronic pain can contribute to depression), so can our psychological health affect us physically (e.g. anxiety can contribute to feelings of chest pain). It is thus critically important to pay attention to the emotional and psychological symptoms associated with all lysosomal storage diseases, including Morquio, and expand our treatment standard of care to include mental health treatment, if necessary.

The first step in understanding and treating psychological conditions in Morquio disease is determining the natural occurrence of psychological symptoms in this population in comparison with non-medical populations. As little has been done in this regard, a pilot study documenting the occurrence rate of psychological issues and overall quality of life in patients with Morquio is the first item in order and will be the focus of this study.

Approximately 20 patients with Morquio disease will be invited to participate, recruited through Emory's Lysosomal Storage Disease Center, as well as through attendance at Morquio support groups and relevant regional, national and/or international meetings. Once consented, patients will be asked to complete three different self-report questionnaires, including the Achenbach System of Empirically Based Assessment (ASEBA) Adult Self-Report (ASR) or Older Adult Self-Report (OASR) questionnaire, the Short Form 36-item Health Questionnaire (SF-36), and the Brief Pain Inventory (BPI). Group aggregate data only will be reported; individual questionnaire content and results will be held confidential, except as in accordance with Georgia law relating to reporting of child or elder abuse, suicidal and/or homicidal intent. Completion of these questionnaires will complete subjects' participation in this pilot study.

ELIGIBILITY:
Inclusion Criteria:

1. Documented clinical diagnosis of MPS IVA based on clinical signs and symptoms of MPS IVA and documented reduced fibroblast or leukocyte GALNS enzyme activity or genetic testing confirming diagnosis of MPS IVA.
2. Subject is at least 18 years old.
3. Subject must provide informed consent prior to study participation.
4. Subject was a participant in the MAP study (Phase I) and is now receiving (or plans to receive in the near future) enzyme replacement therapy in the EAP or commercial setting. If receiving ERT for the treatment of Morquio A syndrome, subject has been on treatment for less than 1 year.

   -or-
5. Subject was not enrolled in the MAP study, but plans to start receiving ERT for Morquio A syndrome in the near future and is willing to take all baseline questionnaires which were included in MAP, prior to beginning ERT for Morquio A syndrome .

Exclusion Criteria:

* 1. Previous treatment with ERT prior to participation in phase 1(MAP).

  2. Previous hematopoietic stem-cell transplant

  3. Patient has a clinically significant disease (with the exception of symptoms of Morquio A syndrome), including clinically significant cardiovascular, hepatic, immunologic, pulmonary, neurologic, or renal disease, or other medical condition, serious intercurrent illness, or extenuating circumstances that, in the opinion of the investigator, would confound the effects of Morquio A syndrome upon study variables.

  4. Any condition that, in the view of the Investigator, places the patient at high risk of poor compliance or of not completing the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Morquio A syndrome
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-03; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
ASEBA Self-Report | Every 6 months for 2 years
  Self-report questionnaire assessing psychological and adaptive functioning

SECONDARY OUTCOMES:
Brief Pain Inventory | Every 6 months for 2 years
  Self-report measure of subjective pain levels and interference of pain in daily functioning
SF-36 | Every 6 months for 2 years
  Brief self-report measure of quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Ali, Ph.D., Principal Investigator — Emory University
Locations (1):
- Emory University, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers